CLINICAL TRIAL: NCT00192088
Title: Open-Label Single-Arm Phase II Study of ALIMTA in Combination With Oxaliplatin as First-Line Therapy in Advanced Gastric Carcinoma
Brief Title: A Study of Pemetrexed Plus Oxaliplatin as First Line Therapy in Advanced Gastric Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8059; H3E-IT-S043
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Advanced Gastric Carcinoma
MeSH Terms: interventions — Pemetrexed; Oxaliplatin

INTERVENTIONS:
Drug: pemetrexed
Drug: oxaliplatin

SUMMARY:
Open label single arm phase II study of Pemetrexed plus Oxaliplatin in patients with advanced gastric carcinoma not previously treated with palliative chemotherapy. 43 Patients will be enrolled in this local trial. The primary objective of this study is to determine the response rate of the treatment.Schedule for this study is as follows: 6 cycles/21 days of Pemetrexed 500 mg/m2 followed by Oxaliplatin 120 mg/m2. This study will also include pharmacogenomic and pharmacogenetic investigations in order to assess determinants of efficacy and toxicity of the treatment with Pemetrexed and Oxaliplatin in the study population.

ELIGIBILITY:
Inclusion Criteria

* Histologically proven diagnosis of adenocarcinoma of the stomach (including adenocarcinoma of the gastroesophageal junction)
* Stage IIIB or Stage IV disease, according to American Joint Committee on Cancer criteria, not amenable to curative surgery or radiation
* Disease status must be that of at least of one measurable disease as defined by RECIST criteria.
* Performance Status of 2 on the ECOG Scale.
* Adequate organ function including the following:
* Bone marrow: absolute neutrophil count (ANC) >or equal to 1.5 * 109/L, platelets >or equal to 100 *109/L, hemoglobin > or equal to 10 g/dL.
* Hepatic: bilirubin < or equal to 1.5 x ULN; alkaline phosphatase, aspartate transaminase (AST) and alanine transaminase (ALT) < or equal to 3 x ULN (alkaline phosphatase, AST, ALT minor or equal to 5 x ULN is acceptable if liver has tumor involvement), serum albumin > or equal to3g/dL.
* Renal: Calculated creatinine clearance major or equal to 45 ml/min (using the standard Cockcroft-Gault formula).

Exclusion Criteria

* No Prior palliative chemotherapy for advanced disease
* Previous radiation therapy is allowed but should have been limited and must not have included whole pelvis radiation. Patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed at least 30 days before study enrollment
* Known or suspected brain metastasis
* Second primary malignancy (except for in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or other malignancy treated at least 5 years previously with no evidence of recurrence)
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of pemetrexed plus oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2004-05; Study Completion 2006-05

PRIMARY OUTCOMES:
The primary objective of this study is to determine the response rate of Pemetrexed plus oxaliplatin as first-line therapy in patients with advanced gastric carcinoma.

SECONDARY OUTCOMES:
The secondary objectives of this study are to evaluate:
The following time to event efficacy measures:Duration of overall response for responding patients-Time to documented progressive disease-Time to treatment failure-Overall survival-The quantitative and qualitative toxicity of pemetrexed plus oxaliplatin.
Determinants of efficacy and toxicity of the treatment with pemetrexed and oxaliplatin in the patient population by means of pharmacogenomic and pharmacogenetics investigations: Quantitative analysis of TS, DHFR, GARFT, RFC, MRP5, DPD, TP, FPGS and ERCC1

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Monday-Friday 9 am-5 pm Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (13):
- Italy (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ancona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brescia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gorgonzola
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mantova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varese
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-371-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verona